CLINICAL TRIAL: NCT03378947
Title: EBV-associated Diffuse Large B Cell Lymphoma NOS in Non Immunocompromised Patients : a French Retrospective Case Study
Brief Title: EBV-associated Diffuse Large B Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Hospices civils de lyon
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: To Characterize and Compare Clinical, Pathological and Molecular Features
Keywords: EBV, DLBCL
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical and pathological data EBV-related GZL and DLBCL — Invesrigators will retrospectively collect clinical and pathological data of all EBV-related GZL and DLBCL in immunocompetent patients diagnosed in the pathology department Centre Hospitalier Lyon Sud.
  Investigators will analyze their clinical feature and prognosis.

SUMMARY:
The aim of this study is to characterize and compare clinical, pathological (histology, immunophenotype) and molecular features of EBV-related GZL and DLBCL: do they belong to the same entity or to two different subtypes of EBV-related lymphoma ?

DETAILED DESCRIPTION:
Recent progresses in the understanding of lymphoma biology allowed the identification of new categories in the WHO classification of lymphoid neoplasm. Among these new entities, grey zone lymphoma (GZL) between classical Hodgkin lymphoma and diffuse large B cell lymphoma entered the classification as a provisional entity in 2008 and Diffuse large B cell lymphoma (DLBCL) EBV-associated not otherwise specified in patient without history of immunodepression in 2016. These entities need however to be further characterized as no clear pathological definition and distinction between EBV related GZL and EBV related DLBCL are proposed in the literature.

After primary infection that occurs in almost 80% of young adult population in western country, EBV latency state settles in a small portion of B cells. The virus is known to promote B-cells proliferation and transformation through complex mechanisms.

EBV-associated lymphoproliferative disorders have already been largely studied in immunocompromised host (human immunodeficiency virus, congenital immunodeficiency, immunosuppressor and post-transplant lymphoproliferative disorder, e.g.), but its role is largely unknown in patients with no history of immunodeficiency. Whether these patients arbor an underlying type of immune deficiency has not yet been established, even though immunosenecence in elderly or immaturity of the immune system in children has been postulated in those population.

Based on former definition, EBV-associated lymphoproliferation were usually the apanage of classical Hodgkin lymphoma (cHL) or immunodeficiency-associated lymphoproliferative disorders. However, as published recently, several different histological patterns with intermediate features between primary mediastinal B cell lymphoma (PMBCL) and classical Hodgkin lymphoma (cHL), namely grey zone lymphoma (GZL), but also diffuse large B cell lymphoma (DLBCL) were described to be EBV-associated. On the clinical point of view, patients with GZL are young and have a poor prognosis. Data regarding EBV+ DLBCL are discordant and further studies are warranted, even though initial report concluded to a poor prognosis for these patients.

ELIGIBILITY:
Inclusion Criteria:

* all EBV-related GZL and DLBCL in immunocompetent patients
* Age minimum: 18 years old

Exclusion Criteria:

* Another diagnosis than EBV-related GZL and DLBCL
* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will retrospectively collect clinical and pathological data of all EBV-related GZL and DLBCL in immunocompetent patients diagnosed in the pathology department Centre Hospitalier Lyon Sud since 2000.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
status at last follow up | up to 48 months
  Investigators will retrospectively collect clinical and pathological data of all EBV-related GZL and DLBCL in immunocompetent patients diagnosed in the pathology department Centre Hospitalier Lyon Sud.- Clinical data will be extracted from medical records, outcome and status at last follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- HCL, Lyon, Pierre Bénite, France